CLINICAL TRIAL: NCT06466070
Title: The Role of Robotic Surgery in Pulmonary Metastasectomy: a Retrospective Multicenter Study
Brief Title: Robotic Surgery in Pulmonary Metastasectomy
Acronym: ROME
Status: Enrolling by invitation | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Collaborators: Istituto Europeo di Oncologia (Other); Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Stefano Viscardi, MD, Scientific Institute San Raffaele
Other Study IDs: CE: 23/INT/2023
Record Dates: First submitted 2024-05-29; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Primary Solid Tumors
Keywords: pulmonary metastasectomy; robot-assisted thoracoscopic surgery; video-assisted thoracoscopic surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- open (thoracotomy): Nowadays, pulmonary metastasectomy is performed in RATS, VATS or thoracotomy. A thoracotomy is a surgical procedure during which a surgeon accesses the lungs and other nearby organs through an incision in the chest wall.
- RATS (robot-assisted thoracoscopic surgery): RATS is a minimally invasive surgical technique allowing enhanced view, accurate and complex movements, and high ergonomics for the surgeon.
- VATS (video-assisted thoracoscopic surgery): VATS is minimally invasive thoracic surgery that does not use a formal thoracotomy incision.

SUMMARY:
The study is observational, multicenter retrospective and will involve multiple research centers. The aim is to outline the indications for surgical management with robot-assisted pulmonary metastasectomy through a confrontation of robot-assisted thoracoscopic surgery (RATS) with video-assisted thoracoscopic surgery (VATS) and thoracotomy. The study will focus on pulmonary metastasectomies from any primary solid tumor (with the exception of lung cancer). There are no risks for the patients, as this is a retrospective data collection.

DETAILED DESCRIPTION:
The investigators will identify selection criteria according to ASA score (American Society of Anaesthesiologists physical status classification system ) and co-morbidities, respiratory function, control and staging of the primary pathology, number and position of metastases. The investigators will assess the robotic approach performance in the different anatomical resections (lobectomies, bilobectomies, segmentectomies,pneumectomies) considering potential intra- and post-operative complications, over than rates of positive margins.

It analyses cases of pulmonary metastasectomy performed with a minimally invasive approach such as robot-assisted thoracoscopic surgery (RATS) and video-assisted thoracoscopic surgery (VATS), or with a traditional open approach. More precisely, it will compare RATS vs VATS as well as RATS vs open.

It was decided to exclude simple wedge resections since, in light of the minimal resection of parenchyma and the costs sustained for the equipment, they are preferably carried out by VATS.

Criteria for the inclusion of patients:

1. The patient can be candidate in terms of ASA score, cardiac, kidney, liver and respiratory function
2. The primary pathology is under control or controllable
3. Absence of extrapulmonary metastases that are not controlled or controllable

Exclusion criteria:

* Age >/=; then 18 years at the moment of surgery
* Patients who cannot undergo surgery, as they do not meet the conditions outlined above.

ELIGIBILITY:
Inclusion Criteria:

* The patient can be candidate in terms of ASA score, cardiac, kidney, liver and respiratory function
* The primary pathology is under control or controllable
* Absence of extrapulmonary metastases that are not controlled or controllable

Exclusion Criteria:

* Age >/= ; then 18 years at the moment of surgery
* Patients who cannot undergo surgery, as they do not meet the conditions outlined above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will focus on pulmonary metastasectomies from any primary solid tumor (with the exception of lung cancer). The anatomical resections considered will be segmentectomy, lobectomy, bilobectomy and pneumonectomy. It was decided to exclude simple wedge resections since, in light of the minimal resection of parenchyma and the costs sustained for the equipment, they are preferably carried out by VATS.
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PERIOPERATIVE OUTCOME | from hospitalization to the discharge date at maximum one week
  The primary objective consists in the definition of indication of the robotic approach in pulmonary metastasectomy.
  The investigators will measure the potential technical superiority of Robotic Assisted Thoracoscopic Surgery (RATS), as compared to Video Assisted Thoracic Surgery (VATS) and thoracotomy, in the different types of anatomical resection for lung metastasectomy, by analizing intra- and post-operative complications, which will be categorized according to Clavien-Dindo scale.
PERIOPERATIVE OUTCOME 2 | from surgery to time of pathological response
  The primary objective consists in the definition of indication of the robotic approach in pulmonary metastasectomy.
  The investigators will measure the potential technical superiority of Robotic Assisted Thoracoscopic Surgery (RATS), as compared to Video Assisted Thoracic Surgery (VATS) and thoracotomy, in the different types of anatomical resection for lung metastasectomy, by analizing the rate of resection radicality.

SECONDARY OUTCOMES:
PATHOLOGICAL OUTCOME | from surgery to time of pathological response
  The investigators will measure the impact of the robotic approach on lymphadenectomy comparing the cases from the Robotic Assisted Thoracic Surgery (RATS) group with the ones from Video Assisted Thoracic Surgery (VATS) and open group, by analizing the number of cases which underwent radical lymphnode dissection or lymphnode sampling.
PATHOLOGICAL OUTCOME 2 | from surgery to time of pathological response
  The investigators will measure the impact of the robotic approach on lymphadenectomy comparing the cases from the Robotic Assisted Thoracic Surgery (RATS) group with the ones from Video Assisted Thoracic Surgery (VATS) and open group, by analizing the number of resected hilar and mediastinal lymphnodes.
PATHOLOGICAL OUTCOME 3 | from surgery to time of pathological response
  The investigators will measure the impact of the robotic approach on lymphadenectomy comparing the cases from the Robotic Assisted Thoracic Surgery (RATS) group with the ones from Video Assisted Thoracic Surgery (VATS) and open group, by analizing the frequency of positive lymphnodes.
PATHOLOGICAL OUTCOME 4 | from surgery to time of pathological response
  The investigators will measure the impact of the robotic approach on lymphadenectomy comparing the cases from the Robotic Assisted Thoracic Surgery (RATS) group with the ones from Video Assisted Thoracic Surgery (VATS) and open group, by analizing the frequency of unexpected positive lymphnodes.

OTHER OUTCOMES:
ONCOLOGICAL LONG TERM OUTCOME | From the discharge date to the follow up at 1year; 3 years and 5 years
  The investigators will evaluate the potential oncological benefit of Robotic Assisted Thoracic Surgery (RATS) by analizing Overall Survival (OS) of patients subjected to robotic resections, compared to Video Assisted Thoracoscopic Surgery (VATS) and open groups.
ONCOLOGICAL LONG TERM OUTCOME 1 | From the discharge date to the follow up at 1year; 3 years and 5 years
  The investigators will evaluate the potential oncological benefit of Robotic Assisted Thoracic Surgery (RATS) by analizing Disease-Free Interval (DFI) of patients subjected to robotic resections, compared to Video Assisted Thoracoscopic Surgery (VATS) and open groups.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IFO - Istituto Nazionale Tumori Regina Elena di Roma, Rome, Italy / Rome
  - Istituto Europeo di Oncologia, Milan, Italy/Milan
  - Istituto Clinico Humanitas, Rozzano, Italy/Milan